CLINICAL TRIAL: NCT02943174
Title: MIND Programme for Cancer Patients: A Group Intervention Programme Based on Third Wave Psychotherapies
Brief Title: MIND Programme for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Inês A Trindade, PhD, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINEICC-1-IAT; SFRH/BD/101906/2014 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIND Programme for cancer (Experimental): MIND programme for cancer is a manualized acceptance, mindfulness and compassionate-based group intervention for cancer patients. It included 8 weekly group sessions, 2h hours each, run in small groups (ranging from 6 to 12 participants).
  Participants in this group also receive cancer treatment as usually performed at the Coimbra University Hospital.
  Interventions: Behavioral: MIND programme for cancer patients; Other: Treatment as Usual (TAU)
- Treatment as Usual (TAU) (Other): Cancer treatment as usually performed at the Coimbra University Hospital.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: MIND programme for cancer patients — Psychotherapeutic programme based on Acceptance, Mindfulness and Compassion for cancer patients Other: Cancer Treatment as Usual
  Arms: MIND Programme for cancer
Other: Treatment as Usual (TAU) — Standard personalized treatment of cancer

SUMMARY:
This investigation aims to apply and test the acceptability of an acceptance, mindfulness and compassionate-based intervention structured for cancer patients. MIND programme for cancer thus comprises 8 weekly group sessions, lasting 1 and a half hour each, run in small groups at an Oncology Service at the Coimbra's University Hospital. For each week participants have assigned homework (e.g., mindfulness exercises). This programme mainly aims to increase participants' physical and psychosocial quality of life, and attenuate depressed mood and anxiety.

DETAILED DESCRIPTION:
The sample will include diagnosed cancer patients recruited at an Oncology Service at the Coimbra's University Hospital. Patients will be approached by their doctor to assess their level of interest in the investigation. Patients who demonstrate interest will go through a Screening interview conducted by a licensed psychologist that aims explain the structure and arms of the investigation, to collect demographic data, and whether the patient meets the inclusion criteria for the study. Patients who meet the inclusion criteria and demonstrate interest in participating in the study, will sign an informed consent. All ethical requirements for research with humans are guaranteed.

Afterwards, participants will be allocated in two groups (experimental and control group). Both groups will maintain the medical treatment as usual (TAU). Additionally, the experimental group will enroll in the MIND programme for cancer patients, also provided by a licensed psychologist.

Both groups will concurrently complete a protocol of self-report measures and their medical data will be collected by the medical staff of the Hospital.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer (stages I-III)

Exclusion Criteria:

* severe psychopathology
* difficulty in completing self-report measures

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Changes in psychopathology (namely, depression and anxiety symptoms) | From Baseline to follow-up
  Measured by DASS-21
Changes in Quality of Life | From Baseline to follow-up
  Measured by the World Health Organization Quality of Life questionnaire (WHOQOL-BREF)